CLINICAL TRIAL: NCT03844750
Title: A Phase II Study of Preoperative Immunotherapy in Patients With Colorectal Cancer and Resectable Hepatic Metastases
Brief Title: Preoperative Immunotherapy (Pembrolizumab) for Patients With Colorectal Cancer and Resectable Hepatic Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Chloe Atreya, MD, PhD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); MedPacto, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chloe Atreya, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 187015; NCI-2018-03165 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-07; First posted 2019-02-18 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
Keywords: Resectable hepatic metastases; Surgery; Immunotherapy; Adjuvant Treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy; pembrolizumab; vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vactosertib, pembrolizumab, surgery) (Experimental): Neoadjuvant pembrolizumab will be administered at a fixed dose of 200 mg (IV) for 1 cycle plus 200 mg vactosertib (PO QD, 5 days per week x 2 weeks). Adjuvant pembrolizumab (400 mg IV) + vactosertib (200 mg PO QD Cycle 1, 5 days per week, Cycles 2 and beyond (200 mg BID, 5 days per week) will be administered for up to eight 6-week cycles
  Interventions: Procedure: Hepatectomy; Biological: Pembrolizumab; Drug: Vactosertib

INTERVENTIONS:
Procedure: Hepatectomy — Undergo liver resection.
  Other Names: Liver Resection
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Vactosertib — Given orally
  Other Names: EW-7197

SUMMARY:
This phase II trials studies how well pembrolizumab and vactosertib work after standard of care chemotherapy in patients with colorectal cancer that has spread to the liver that can be removed by surgery (resectable hepatic metastases). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Vactosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and vactosertib after standard of care chemotherapy, but before liver metastases surgery, may help shrink the cancer prior to surgery. This study also investigates pembrolizumab and vactosertib after liver metastases surgery, decrease the risk of the cancer recurring (coming back).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the change in the populations of tumor infiltrating lymphocytes (TILs) induced by neoadjuvant pembrolizumab plus vactosertib in participants with metastatic colorectal cancer (mCRC).

SECONDARY OBJECTIVES:

I. To establish the safety/toxicity profile of pembrolizumab-based treatment in the perioperative setting for participants with colorectal cancer (CRC) with resectable hepatic metastases.

II. To explore the efficacy of pembrolizumab plus vactosertib in participants with CRC with resectable hepatic metastases.

EXPLORATORY OBJECTIVES:

I. To determine the impact of pembrolizumab-based treatment on programmed death-ligand 1 (PD-L1) expression in tumor cells and tumor-infiltrating immune cells (TIICs), in participants with mCRC.

II. To determine the change in T cell repertoire within the tumor and blood induced by neoadjuvant pembrolizumab-based treatment in participants with mCRC.

III. To explore molecular profiles to identify potentially predictive biomarkers for participants with metastatic CRC treated with immunotherapy (including but not limited to microsatellite instability (MSI) testing).

IV. To correlate change in TIICs, PD-L1 expression, and T cell repertoires as well as molecular profiles with response/resistance and toxicity.

V. To identify immune response messenger ribonucleic acid (mRNA) expression analysis to derive signatures associated with tumor response.

VI. To identify genomic mutations and gene copy aberrations associated with response and resistance to therapy.

VII. To correlate changes in microbiome composition and diversity with diet and lifestyle factors.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and vactosertib orally (PO) once a day (QD) for the first cycle 5 days a week for 2 weeks. Participants then undergo standard of care surgical removal of liver metastases approximately 2 weeks (minimum 1 week) after last dose of vactosertib.

OPTIONAL ADJUVANT TREATMENT: After surgery, eligible participants may also receive pembrolizumab and vactosertib every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants who do not undergo optional adjuvant treatment are followed up at 14 days and then every 90 days for up to 1 year. Participants who undergo optional adjuvant treatment are followed up at 30 days and then every 90 days for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed CRC with liver metastases. In addition to liver metastases, extrahepatic metastases (e.g. pulmonary metastases) may be permitted if all other eligibility criteria are met. Participants are permitted to have primary tumor in situ (Neoadjuvant Arm only).
2. Has received previous oxaliplatin-based chemotherapy.

   a. FOLFOX or capecitabine combined with oxaliplatin (CapeOx) does not need to be a direct lead-in to this study.

   b. If chemotherapy is a direct lead-in to this study, concurrent mAb therapy (bevacizumab, cetuximab, or panitumumab) is acceptable, however the antibody must be omitted from the final cycle of chemotherapy prior to pembrolizumab.
3. Is an appropriate candidate to undergo liver biopsy and resection (+/-ablation) of liver metastases (Neoadjuvant Arm Only).
4. Is willing and able to provide written informed consent/assent for the trial. The participants may also provide consent for Future Biomedical Research. However, may participate in the main trial without participating in Future Biomedical Research.
5. Is >=18 years of age on day of signing informed consent.
6. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the investigator. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions (Neoadjuvant Arm Only).
7. Is willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained after last dose of standard of care lead-in chemotherapy [if applicable] and within 28 days prior to first dose of pembrolizumab (Neoadjuvant Arm Only).
8. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
9. Has adequate organ function within 10 days of treatment initiation.

   - Absolute neutrophil count (ANC) >= 1,500/microliter (uL) (within 10 days of treatment initiation).
   * Platelets >= 100,000/uL (within 10 days of treatment initiation).
   * Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment).
   * Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)) >= 60 mL/min for participants with creatinine levels > 1.5 x institutional ULN (within 10 days of treatment initiation).

     * Creatinine clearance should be calculated per institutional standard.
   * Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation).
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x ULN (within 10 days of treatment initiation).
   * Albumin >= 2.5 mg/dL (within 10 days of treatment initiation).
   * International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation).
   * Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participants is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation).
10. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication (day 1). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
12. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    *Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participants.
13. Have locally confirmed microsatellite stable (MSS) or Mismatch repair proficient (pMMR) Colorectal cancer (CRC). MSS is defined as 0-1 allelic shifts among 3-5 tumor microsatellite loci using a Polymerase chain reaction (PCR)-based assay. pMMR is defined as presence of protein expression of 4 DNA mismatch repair (MMR) enzymes (MLH1, MSH2, MSH6 and PMS2) by immunohistochemistry.
14. Have no radiographic evidence of malignancy as assessed by Investigator (Adjuvant Phase Only).

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

   * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks since the last dose of the previous investigational agent or device use.
2. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
4. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
5. Has active hepatitis B (defined as hepatitis B surface antigen (HBsAg) reactive) or active hepatitis C virus (HCV) (defined as HCV RNA [qualitative] is detected) infection.
6. Has received prior anti-cancer monoclonal antibody (mAb), systemic anticancer therapy other than FOLFOX (including investigational agents), targeted small molecule therapy, or radiation therapy within 14 days prior to the first dose of study treatment (day 1).

   * Note: Participants must have recovered from all adverse events (AEs) due to a previous therapies to =< grade 1 or baseline. Participant with grade 2 neuropathy or alopecia are eligible. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
7. Has received FOLFOX less than 7 days prior to the first dose of study treatment (day 1). Has not recovered (i.e., =< grade 1 or at baseline) from AEs due to FOLFOX chemotherapy.

   * Note: Participants with =< grade 2 neuropathy or alopecia are exceptions to this criterion and may qualify for the study.
8. Has not recovered adequately from toxicity or complications of a surgery or other procedure, per the assessment of the treating investigator.
9. Has received liver-directed therapy such as radiotherapy or yttrium-90 in the past year involving the lesion to be biopsied. (Neoadjuvant Arm only)
10. Has a known additional malignancy that is progressing or has required active treatment within 5 years prior.

    * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression by imaging for at least 4 weeks by repeat imaging [repeat imaging should be performed during the study screening]), clinically stable, and without requirement of steroid treatment for at least 14 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
12. Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator. Anticoagulation that cannot be safely held to perform the liver biopsy is an example of a contraindication to participation.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Has received any prior immunotherapy including anti-PD-1, anti-PD-L1, or anti-PD-L2 or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137). (Neoadjuvant Arm Only).

17. Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or to any of pembrolizumab's excipients.

18. Has received a live or live-attenuated vaccine within 30 days prior to first dose of the trial drug. Administration of killed vaccines are allowed.

19. Has inferior vena cava/cardiac involvement based on imaging. 20. Has had encephalopathy in the last 6 months. Those participants on rifaximin or lactulose to control their encephalopathy are not allowed.

21. Has had a solid organ or hematologic transplant. 22. Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thora- or paracentesis) is eligible.

23. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (>=150/90mmHg), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvulopathy requiting treatment, active interstitial lung disease, or serious chronic gastrointestinal conditions associated with diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Atreya, MD, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with study collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Vactosertib, Pembrolizumab, Surgery): Neoadjuvant pembrolizumab will be administered at a fixed dose of 200 mg (IV) for 1 cycle plus 200 mg vactosertib (PO once a day (QD), 5 days per week x 2 weeks). Adjuvant pembrolizumab (400 mg IV) + vactosertib (200 mg PO QD Cycle 1, 5 days per week, Cycles 2 and beyond (200 mg twice a day (BID), 5 days per week) will be administered for up to eight 6-week cycles
Period: Overall Study
Arm/Group | Treatment (Vactosertib, Pembrolizumab, Surgery)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vactosertib, Pembrolizumab, Surgery)
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  40 - 49 years old | 1
  50 - 59 years old | 4
  60 - 69 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a >= 2-fold Increase in the Tumor-infiltrating Cells Per Unit Area (5 High Power Fields) in Post- Versus Pre Pembrolizumab Treatment Tumor Specimens.
Description: Tumor-infiltrating immune cells (TIICs) will be analyzed by immunohistochemistry (IHC) in pre- and post-pembrolizumab treatment tumor specimens. The proportion of patients with a >= 2-fold increase (from pre- to post-treatment) in the number of TIICs per unit area (5 high power fields) will be calculated.
Time Frame: Up to 2 years
Population: Due to early study termination by the collaborating sponsor, the funds provided by the collaborating sponsor were no longer available to complete the specific analyses detailed in the primary endpoint. No plans currently exist to fund analysis of this endpoint in the future.
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Participants With Treatment-related, Adverse Events
Description: Adverse events (AEs) will be analyzed including but not limited to all AEs, serious (S)AEs, and fatal AEs using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5 for classification. Due to the potential for late toxicities from pembrolizumab, patients will be followed for 1 year after their last dose of pembrolizumab.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 6
proportion of participants | 1.00

3. Secondary Outcome: Proportion of Participants With Events of Clinical Interest (ECIs)
Description: Specific immune-related AEs (irAEs) will be collected and designated as immune-related events of clinical interest (ECIs). The study will use descriptive statistics to report on the safety/toxicity. Due to the potential for late toxicities from pembrolizumab, patients will be followed for 1 year after their last dose of pembrolizumab
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 6
proportion of participants | 0.33

4. Secondary Outcome: Proportion of Participants With Perioperative Complications
Description: The proportion of participants with reported perioperative complications related to study treatment will be reported.
Time Frame: Up to 1 month
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 6
proportion of participants | 0.17

5. Secondary Outcome: Proportion of Participants With an R0 Resection
Description: Participants who undergo surgical resection of liver metastases will be evaluable and the proportion of participants requiring an R0 resection will be reported
Time Frame: Up to 1 month
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 6
proportion of participants | 0.83

6. Secondary Outcome: Proportion of Participants With a Pathologic Response
Description: Participants who undergo surgical resection of liver metastases will be evaluable and the proportion of participants with a pathological tumor response will be reported
Time Frame: Up to 1 year
Population: Only 1 participant underwent partial colectomy at the time of liver resection surgery enabling reliable determination pathological response in the colon primary
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 1
proportion of participants | 0

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the radiographic response as measured from baseline until the day of surgery will be evaluated using RECIST. Participants with a radiographic complete response (CR) or partial response (PR) before surgery will be reported.
Time Frame: Up to the time of surgery, approximately 14 days
Population: Due to funding constraints, the non-standard of care (planned as research-funded) radiological scan originally planned for this short-interval ORR endpoint was not performed. Therefore, no data for ORR between baseline and date of surgery was collected.
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 0

8. Secondary Outcome: Median Relapse-free Survival (RFS)
Description: The time from objective response defined as radiographic evidence of relapse on surveillance CT scans after surgery to progression or death, whichever occurs first, will be used to determine relapse-free survival for participants who received adjuvant vactosertib and pembrolizumab.
Time Frame: Up to 2 years from day of surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (vactosertib, pembrolizumab, surgery)
Number analyzed (Participants) | 4
months | 14.51 [4.44 to NA] — There were insufficient number of events so an upper limit to the confidence interval could not be calculated.

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Vactosertib, Pembrolizumab, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vactosertib, Pembrolizumab, Surgery) (N=6)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vactosertib, Pembrolizumab, Surgery) (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Skin and subcutaneous tissue disorders, Other (Skin and subcutaneous tissue disorders) | 1 (1) — Spontaneous ecchymosis
Thromboembolic event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated earlier than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03844750/Prot_SAP_000.pdf